CLINICAL TRIAL: NCT02390375
Title: Phase 3 Study to Evaluate the Efficacy and Safety of the DW0929 in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DW-0929_P301
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental): DW-0929
  Interventions: Drug: DW-0929
- B (Active Comparator): Rosuvastatin
  Interventions: Drug: DW-0929; Drug: Rosuvastatin

INTERVENTIONS:
Drug: DW-0929 — 5/10mg
Drug: DW-0929 — 10/10mg
Drug: DW-0929 — 20/10mg
Drug: Rosuvastatin — 5mg F/U study: DW-0929 5/10mg
  Arms: B
Drug: Rosuvastatin — 10mg F/U study: DW-0929 10/10mg
  Arms: B
Drug: Rosuvastatin — 20mg F/U study: DW-0929 20/10mg
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the DW0929 in patients with primary hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Adult over 19years
* Patients with primary hypercholesterolemia whose LDL-C level is below 250mg/dL and TG level is below 350mg/dL
* Patients whose LDL-C level is under 'Anti- dyslipidemia drug administration considered standard' of NCEP ATP III(2004)
* Those who voluntarily written consent to participate in this clinical trial

Exclusion Criteria:

* Uncontrolled hypertension
* Severe renal impairment(CrCl<30mL/min)
* Those who have active liver disease and whose ALT, AST levels greater than twice the upper limit of normal
* Serum creatinine > 2.0mg/dL
* Those who have been geunyukbyeong or rhabdomyolysis caused by using statin or have hypersensitivity to ezetimibe
* Combined cyclosporine -treated patients
* HbA1c ≥ 9%
* TSH ≥ 1.5 X ULN
* HIV-positive person
* Congestive heart failure patients classified as NYHA Class III or IV
* Patients with uncontrolled arrhythmias
* Patients who have malignant tumors needed chemotherapy, radiation therapy, etc.
* Blood clotting disorders
* Patients who had a myocardial infarction within 6 months or cardiovascular bypass surgery, patients who have underwent angioplasty
* Patients who had a history of anxiety or severe typical peripheral arterial disease within three months
* Women of childbearing age who don't agree with contraception during this clinical trials
* Pregnant women or nursing mothers
* Those who take the drug in combination taboo
* Who have been treated for another investigational drug within 30 days
* Unsuitable characters in a clinical trial to test self- determination

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
LDL-C level | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Boramae Hospital, Seoul, Dongjak-gu, South Korea